CLINICAL TRIAL: NCT03489369
Title: A Phase 1, Open-Label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Antineoplastic Activity of Sym022 (Anti-LAG-3) in Patients With Advanced Solid Tumor Malignancies or Lymphomas
Brief Title: Sym022 (Anti-LAG-3) in Patients With Advanced Solid Tumor Malignancies or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sym022-01
Record Dates: First submitted 2018-03-26; First posted 2018-04-05 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Cancer; Solid Tumor; Lymphoma
Keywords: Locally advanced/unresectable; Metastatic solid tumor; Lymphoma; Anti-LAG-3; LAG-3; LAG3
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sym022 (Experimental): Sym022 will be administered at up to 4 planned dose levels.
  Interventions: Drug: Sym022

INTERVENTIONS:
Drug: Sym022 — Sym022 is a recombinant, fully human antibody that binds LAG-3 and blocks the LAG-3/major histocompatibility complex class II (MHC-II) interaction, thus allowing for increased T-cell proliferation and cytokine production.
  Other Names: Anti-LAG-3

SUMMARY:
This is the first study to test Sym022 in humans. The primary purpose of this study is to see if Sym022 is safe and tolerable for patients with locally advanced/unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available.

DETAILED DESCRIPTION:
This study will evaluate the preliminary safety, tolerability, and dose-limiting toxicities (DLTs) of Sym022, an anti-lymphocyte activation gene 3 (anti-LAG-3) monoclonal antibody (mAb). The goal is to establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of sequential escalating doses of Sym022 when administered once every 2 weeks (Q2W) by intravenous (IV) infusion to patient cohorts with locally advanced/ unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available. If an MTD is not identified, a maximum administered dose (MAD) will be determined. Sym022 will be given to patients in escalating dose cohorts; each patient will be given one fixed dose level.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age at the time of obtaining informed consent.
* Documented (histologically- or cytologically-proven) solid tumor malignancy that is locally advanced or metastatic; patients with documented lymphomas.
* Malignancy (solid tumor or lymphoma) that is currently not amenable to surgical intervention due to either medical contraindications or nonresectability of the tumor.
* Refractory to or intolerant of existing therapy(ies) known to provide clinical benefit.
* Measurable or non-measurable disease according to RECIST v1.1 or RECIL 2017.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Not of childbearing potential or who agree to use a highly effective method of contraception during the study beginning within 2 weeks prior to the first dose and continuing until 6 months after the last dose of study drug.

Exclusion Criteria:

* Women who are pregnant or lactating, or intending to become pregnant before, during, or within 6 months after the last dose of study drug. Women of childbearing potential (WOCBP) and fertile men with WOCBP partner(s), not using and not willing to use a highly effective method of contraception.
* Known, untreated central nervous system (CNS) or leptomeningeal metastases, or spinal cord compression, patients with any of the above not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
* Hematologic malignancies other than lymphomas.
* Active thrombosis, or a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 4 weeks prior to Cycle 1/Day 1 (C1/D1) unless adequately treated and considered stable
* Active uncontrolled bleeding or a known bleeding diathesis
* Clinically significant cardiovascular disease or condition
* Significant pulmonary disease or condition
* Current or recent (within 6 months) significant gastrointestinal (GI) disease or condition.
* An active, known, or suspected autoimmune disease, or a documented history of autoimmune disease or syndrome, requiring systemic steroids or other immunosuppressive medications.
* History of organ transplantation (e.g. stem cell or solid organ transplant)
* History of significant toxicities associated with previous administration of immune checkpoint inhibitors that necessitated permanent discontinuation of that therapy
* Patients with unresolved > Grade 1 toxicity associated with any prior antineoplastic therapy, with exceptions.
* Inadequate recovery from any prior surgical procedure, or having undergone any major surgical procedure within 4 weeks prior to C1/D1.
* Known history of human immunodeficiency virus (HIV) or known active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Other Inhibitors of LAG-3
* Any antineoplastic agent for the primary malignancy (standard or investigational) without delayed toxicity within 4 weeks or 5 plasma half-lives, whichever is shortest, prior to first administration of study drug and during study
* Any other investigational treatments within 4 weeks prior to and during study
* Radiotherapy for target lesions within 4 weeks prior to first administration of study drug unless PD has been documented in the lesion following treatment, and during study.
* Radiotherapy for non-target lesions within 1 week prior to first administration of study drug
* Immunosuppressive or systemic hormonal therapy
* Prophylactic use of hematopoietic growth factors within 1 week prior to first administration of study drug and during Cycle 1 of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, FRCPC, Principal Investigator — Princess Margaret Cancer Centre
Locations (3):
- United States (2):
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 0.3 mg/kg dosing of Sym022 every second week (Q2W)
- Dose Level 2: 1.0 mg/kg dosing of Sym022 every second week (Q2W)
- Dose Level 3: 3 mg/kg dosing of Sym022 every second week (Q2W)
- Dose Level 4: 10.0 mg/kg dosing of Sym022 every second week (Q2W)
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 3 | 3 | 3 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 6
Not completed — Documented Progressive Disease | 3 | 2 | 3 | 6
Not completed — Clinical Progression (Worsening of Clini | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.82) | 69 (1.73) | 70.3 (13.28) | 64.8 (6.11) | 65.4 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 4 | 7
  Male | 2 | 2 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 2 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 3 | 3 | 2 | 4 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
ECOG PS [Count of Participants; unit: Participants] — ECOG: Eastern Cooperative Oncology Group PS: Performance status is a measure of how well a person is able to carry on ordinary daily activities while living with cancer, and provides an estimate of what treatments a person may tolerate. It has scores ranging from 0 to 5 with 0 being best and 5 being worst. ECOG is commonly used as a prognostic tool, as a selection criterion for cancer research, and to help determine treatment
  Participants
    0 | 0 | 0 | 1 | 0 | 1
    1 | 3 | 3 | 2 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Treatment Related Adverse Events (AEs).
Description: Assess the safety, tolerability and dose-limiting toxicities of Sym022 on a Q2W schedule to establish the MTD and/or RP2D.
Time Frame: 19 months
Population: Patients evaluable for Maximum Tolerated Dose
Measure: Number; unit: Patients with any DLT
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
Patients with any DLT | 0 | 0 | 0 | 1

2. Secondary Outcome: Evaluation of the Immunogenicity of Sym022.
Description: Serum sampling and incidence (%) per dose level to assess the potential for anti-drug antibody (ADA) formation. Count of participants show the number of participants who were tested positive for anti-Sym022 ADA.
Time Frame: 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 1 | 0 | 0 | 0

3. Secondary Outcome: Evaluation of Objective Response (OR) or Stable Disease (SD).
Description: Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), Response Evaluation Criteria in Lymphomas 2017 (RECIL 2017), or Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST), depending on tumor type. The numbers shown below correspond to the values related to RECIST v1.1.
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 0 | 1 | 0

4. Secondary Outcome: Time to Progression (TTP) of Disease.
Description: Based on time of enrollment to first evidence of progression on imaging studies, as assessed by RECIST v1.1, RECIL 2017, or iRECIST, depending on tumor type. The numbers shown below correspond to the values related to RECIST v1.1.
Time Frame: 13 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
months | 1.64 [1.6 to 3.0] | 5.59 [1.7 to 5.6] | 6.14 [1.6 to 9.3] | 1.58 [0.7 to 3.6]

5. Secondary Outcome: Area Under the Concentration-time Curve in a Dosing Interval (AUC).
Description: Will be estimated using non-compartmental methods and actual timepoints.
Time Frame: 19 months
Measure: Mean (Standard Deviation); unit: hours*μg/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
hours*μg/mL | 926 (151) | 3860 (1010) | 10000 (1720) | 28300 (7110)

6. Secondary Outcome: Maximum Concentration (Cmax)
Description: Will be derived from observed data.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours as administered Q2W (every second week)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
μg/mL | 7.61 (1.706) | 29.58 (4.060) | 76.54 (4.865) | 243.99 (88.517)

7. Secondary Outcome: Time to Reach Maximum Concentration (Tmax)
Description: Will be derived from observed data.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours as administered Q2W (every second week)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
hours | 3.06 (2.018) | 4.52 (2.869) | 2.43 (2.271) | 1.98 (1.636)

8. Secondary Outcome: Trough Concentration (Ctrough)
Description: Will be derived from observed data.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours as administered Q2W (every second week)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 6
μg/mL | 0.85 (0.465) | 4.09 (1.931) | 12.22 (1.547) | 44.10 (12.475)

9. Secondary Outcome: Terminal Elimination Half-life (T½)
Description: Will be estimated using non-compartmental methods and actual timepoints.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours as administered Q2W (every second week)
Population: For some participants in "Dose Level 4", the time span between the first and the last data point for the terminal rate constant did not cover at least 1.5 halflives, and these participants are therefore not part of the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
hours | 119.48 (33.674) | 133.12 (35.491) | 152.94 (24.570) | 169.05 (18.830)

10. Secondary Outcome: Clearance (CL)
Description: Will be estimated using non-compartmental methods and actual timepoints.
Time Frame: 0, 2, 4, 8, 24, 48, 168 hours and 336 hours as administered Q2W (every second week)
Population: Participants with an extrapolated AUC above 20% (for single dose administration) are not part of the analysis.
Measure: Mean (Standard Deviation); unit: (mL/h)/kg
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 2 | 1 | 2 | 0
(mL/h)/kg | 0.32 (0.006) | 0.31 (NA) — Standard Deviation is not available since the overall number of participants analyzed is 1 | 0.24 (0.060) |

ADVERSE EVENTS:
Time Frame: From signing of informed consent through 30 days after last dose; through 2 months (or 4 months to 2 years) follow-up if related critical AEs persist
Description: Only treatment-emergent adverse events are presented in clinicaltrials.gov
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 5/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=6)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 2 (4) | 1 (1) | 1 (4)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical discharge (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT03489369/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT03489369/SAP_001.pdf